CLINICAL TRIAL: NCT00685438
Title: Observational Study of Skin Erythema by Spectrophotometer, and UV Exposure With Viospore Ultraviolet Monitors at Extreme Altitude (Mt. Everest, North Side)
Brief Title: Ultraviolet Exposure, Antioxidant Use and Skin Erythema at Extreme High Altitude
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Ontario Centres of Excellence (Industry)
Responsible Party: Ivy Cheng, Sunnybrook Health Sciences Center
Other Study IDs: 005-2007
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Altitude; Ultraviolet Rays; Antioxidants; Oxidative Stress; Erythema
Keywords: Environmental Medicine; Altitude; Ultraviolet Rays; Antioxidants; Oxidative Stress; Erythema
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
With the increasing tourism and adventure travel into extreme environments comes the need to reassess the required protection against ultraviolet (UV) radiation and possible other oxidative stresses. This is an observational study of UV radiation exposure and skin erythema while at extreme altitude (Mt. Everest). In addition to UV exposure, skin erythema, antioxidant use (such as vitamins C and E) will be measured.

Hypothesis:

1. UV radiation at extreme altitude has larger effects on the skin than at sea level; therefore requiring an adjustment of the antioxidant use for adequate protection.
2. The skin is an accurate reflection of UV and oxidative stress exposure
3. The efficacy of oxidatives stress is reflective of the ethnicity of the individual.

DETAILED DESCRIPTION:
The literature widely acknowledges the deleterious effects of UV radiation on skin health, via production of oxidative free radicals. Consequently, there have been numerous studies on the potential dermatological/anti-carcinogenic benefits of anti-oxidants, such as vitamins C and E, melatonin, green tea, zinc, and selenium. There is, however, a limited amount of literature on the quantity of UV exposure in high-risk settings, such as extreme altitude and equatorial zones. Currently, there is no literature on UV exposure on Mount Everest. Additionally, the efficacy of antioxidants (topical or systemic) has not yet been established in this environment.

This will be an observational study where the principal investigator will collect accumulated ultraviolet exposure at different extreme altitudes during a 6 week period of a summit expedition on the north side of Mt. Everest. Included in the data collection will be patient demographics, time, altitude, temperature, use of anti-oxidants, sunscreen (weighed), and skin erythema (spectophotometer).

ELIGIBILITY:
Inclusion Criteria:

* Participants part of the expedition who are willing to wear the monitor, and disclose information of diet/antioxidant supplements and topical sunblock.

Exclusion Criteria:

* Participants who are unwilling to carry the UV monitor or disclose their demographics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 9 Mountaineers with intention to summit Everest (1 American, 1 British, 1 German, 5 Australians, 1 Asian-Australian) 4 Trekkers with intention to go to 7000m (2 Americans, 1 Asian, 1 British) 12 climbing sherpas (11 Nepali and 1 Tibetan)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-04; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivy S Cheng, MD, Principal Investigator — Sunnybrook Hospital Emergency Department; Lothar D Lilge, PhD, Principal Investigator — Ontario Cancer Institute
Locations (1):
- Mount Everest, North side, Kathmandu, Nepal

REFERENCES:
- [Background] Solar and ultraviolet radiation. IARC Monogr Eval Carcinog Risks Hum. 1992;55:1-316. No abstract available. PMID 1345607
- [Background] Nishigori C. Cellular aspects of photocarcinogenesis. Photochem Photobiol Sci. 2006 Feb;5(2):208-14. doi: 10.1039/b507471a. Epub 2005 Dec 1. PMID 16465307
- [Background] Pinnell SR. Cutaneous photodamage, oxidative stress, and topical antioxidant protection. J Am Acad Dermatol. 2003 Jan;48(1):1-19; quiz 20-2. doi: 10.1067/mjd.2003.16. PMID 12522365
- [Background] Moehrle M, Dennenmoser B, Garbe C. Continuous long-term monitoring of UV radiation in professional mountain guides reveals extremely high exposure. Int J Cancer. 2003 Mar 1;103(6):775-8. doi: 10.1002/ijc.10884. PMID 12516097
- [Background] Solorzano et al. Columbia: 40 Million People Exposed to Extreme Ultraviolet Radiation During the Whole Year. Radiation Protection Dosimetry 2000; 91(1-3): 325-328
- [Background] Moehrle M, Garbe C. Does mountaineering increase the incidence of cutaneous melanoma? A hypothesis based on cancer registry data. Dermatology. 1999;199(3):201-3. doi: 10.1159/000018274. PMID 10592397
- [Background] Bartsch P, Bailey DM, Berger MM, Knauth M, Baumgartner RW. Acute mountain sickness: controversies and advances. High Alt Med Biol. 2004 Summer;5(2):110-24. doi: 10.1089/1527029041352108. PMID 15265333
- [Background] Bailey DM, Kleger GR, Holzgraefe M, Ballmer PE, Bartsch P. Pathophysiological significance of peroxidative stress, neuronal damage, and membrane permeability in acute mountain sickness. J Appl Physiol (1985). 2004 Apr;96(4):1459-63. doi: 10.1152/japplphysiol.00704.2003. Epub 2003 Oct 31. PMID 14594861
- [Background] Moehrle M, Garbe C. Personal UV dosimetry by Bacillus subtilis spore films. Dermatology. 2000;200(1):1-5. doi: 10.1159/000018306. PMID 10681605
- [Derived] Cheng I, Kiss A, Lilge L. An observational study of personal ultraviolet dosimetry and acute diffuse reflectance skin changes at extreme altitude. Wilderness Environ Med. 2013 Dec;24(4):390-6. doi: 10.1016/j.wem.2013.05.007. Epub 2013 Sep 25. PMID 24075057
- See also: Ultraviolet monitors being used — http://www.biosense.de/hope-e.htm